CLINICAL TRIAL: NCT00565877
Title: A Randomized, Controlled Trial Evaluating Post-Insertion Neck Ultrasound in Peripherally Inserted Central Catheter Procedures
Brief Title: The Application of Neck Ultrasound in the Assessment of Peripherally Inserted Central Catheter (PICC) Tip Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 13466A
Record Dates: First submitted 2007-11-29; First posted 2007-11-30 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Peripherally Inserted Central Catheter Insertion Technique
Keywords: Catheter; Peripherally inserted central catheter; ultrasound; malposition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 - Neck Ultrasound (Experimental): post-PICC insertion ultrasound inspection of the ipsilateral neck
  Interventions: Other: Ultrasound inspection
- 2 - Control (No Intervention): No post-PICC insertion ultrasound inspection of the ipsilateral neck

INTERVENTIONS:
Other: Ultrasound inspection — post-PICC insertion Ultrasound inspection of the ipsilateral neck for PICC in a malposition (ipsilateral internal jugular vein)
  Arms: 1 - Neck Ultrasound

SUMMARY:
Insertion of peripherally inserted central catheters (PICCs) at the bedside may result in tip malposition. This study was designed to evaluate whether the addition of ultrasound (US) inspection of the ipsilateral neck provides immediate recognition of PICCs in aberrant position facilitating catheter reposition prior to completion of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 years old) ordered for a peripherally inserted central catheter insertion

Exclusion Criteria:

* patients unable to provide informed consent
* previous peripheral inserted central catheter placement at the institution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2004-10; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Rate of PICCs in the ipsilateral internal jugular vein malposition as detected by post-procedure chest x-ray | Same day

SECONDARY OUTCOMES:
Duration of PICC procedure. | Same day.

CONTACTS AND LOCATIONS:
Overall Officials: John P Kress, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States